CLINICAL TRIAL: NCT03930121
Title: Transcranial Direct Current Stimulation to Enhance Training Effectiveness in Chronic Post-Stroke Aphasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DC-Train-Aphasia
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Aphasia; Post-stroke
Keywords: Rehabilitation; Intensive speech-language therapy; Transcranial direct current stimulation
MeSH Terms: conditions — Aphasia | interventions — Transcranial Direct Current Stimulation; Speech Therapy

STUDY DESIGN:
Intervention Model Description: Two daily sessions of intensive speech-language therapy combined with transcranial direct current stimulation of the left primary motor cortex (M1)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Anodal transcranial direct current stimulation (tDCS) combined with speech-language therapy (SLT, including naming therapy and communicative-pragmatic therapy)
  Interventions: Other: Anodal transcranial direct current stimulation (tDCS) combined with speech-language therapy (SLT, including naming therapy and communicative-pragmatic therapy)
- Control group (Sham Comparator): Placebo stimulation (using sham-tDCS) combined with SLT
  Interventions: Other: Anodal transcranial direct current stimulation (tDCS) combined with speech-language therapy (SLT, including naming therapy and communicative-pragmatic therapy)

INTERVENTIONS:
Other: Anodal transcranial direct current stimulation (tDCS) combined with speech-language therapy (SLT, including naming therapy and communicative-pragmatic therapy) — Two daily sessions of intensive SLT combined with tDCS of the left primary motor cortex (M1)

SUMMARY:
The aim of the study is to investigate whether intensive speech-language therapy (SLT) combined with anodal transcranial direct current stimulation (tDCS) leads to better communication performance than SLT combined with placebo stimulation (using sham-tDCS).

DETAILED DESCRIPTION:
Intensive speech-language therapy (SLT) can promote recovery from chronic post-stroke aphasia, but effect sizes are moderate. This highlights the pressing need to explore adjunct strategies, such as transcranial direct current stimulation (tDCS), to enhance training effectiveness. Recently, the investigators provided evidence from a single-center randomized controlled trial (RCT) suggesting that anodal-tDCS of the left primary motor cortex (M1) improves naming and communication ability in chronic post-stroke aphasia, with medium-to-large effect sizes. However, prior to integration into clinical routine, a multi-center RCT with adequate power, duration, and outcomes relevant to everyday life is required, which is the goal of the present study. After trial completion, a workshop with relevant stakeholders will ensure transfer into best-practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* left-hemisphere cortical or subcortical stroke with first-ever aphasic symptoms
* at least 6 months post-onset of stroke;
* aphasia, as determined by the Aachen Aphasia Test (AAT);
* 13 moderate-to-severe word finding difficulties (maximum of 75% correct items on a computerized naming task at baseline);
* at least 1 correct reaction on the first part of the AAT subscale Token Test (ensuring basic comprehension skills);
* at least 1 point on the communicative task of the AAT subscale Spontaneous Speech (ensuring basic communication abilities);
* German as first language;
* intact left-hemisphere "hand knob" without right prefrontal lesions for placement of tDCS electrodes, as confirmed by magnetic resonance imaging or computer tomography scans.

Exclusion Criteria:

* contraindications for tDCS (e.g., cardiac pacemaker, history of seizures, implanted metal inside the head);
* more than one clinically apparent stroke with aphasic symptoms;
* other severe neurological diseases (e.g., brain tumor, and subdural hematoma);
* epilepsy with seizures during the last 12 months prior to study start and/or intake of sedating antiepileptic drugs (barbiturates and benzodiazepines),
* history of severe alcohol or drug abuse;
* current severe depression;
* current psychosis or other relevant psychiatric condition;
* very severe apraxia of speech, as revealed by Hierarchical Word Lists;
* severe non-verbal cognitive deficits, as indicated by the Corsi Block-Tapping Task;
* severe uncontrolled medical problems;
* severely impaired vision or hearing that prevents patients from engaging in intensive SLT;
* changes in centrally active drugs within 2 weeks prior to study inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Change in communication ability, as assessed by the Amsterdam Nijmegen Everyday Language Test | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  Amsterdam Nijmegen Everyday Language Test (A-scale; parallel versions used in counterbalanced order across participants); cf. Blomert L, Kean ML, Koster C, et al. Amsterdam-Nijmegen Everyday Language Test-Construction, Reliability and Validity. Aphasiology 1994; 8: 381-407.

SECONDARY OUTCOMES:
Change in naming ability, as assessed based on personally relevant trained and untrained items, consistent with previous work (see description) | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  Personally relevant trained and untrained items, consistent with previous work; cf. Meinzer M, Darkow R, Lindenberg R, et al. Electrical stimulation of the motor cortex enhances treatment outcome in post-stroke aphasia. Brain 2016; 139: 1152-1163.
Change in (non-)verbal communication, as assessed by the Scenario Test | Before the 3-week treatment period; 6-month follow-up
  Scenario Test; cf. Nobis-Bosch R, Abel S, Krzok F, et al. Szenario Test-Testung verbaler und nonverbaler Aspekte aphasischer Kommunikation. ProLog, in preparation.
Change in (non-)verbal communication, as assessed by the Communicative Effectiveness Index | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  Communicative Effectiveness Index; cf. Lomas J, Pickard L, Bester S, et al. The Communicative Effectiveness Index: development and psychometric evaluation of a functional communication measure for adult aphasia. J Speech Hear Disord 1989; 54: 113-124.
Change in attention and executive function, as assessed by the subscales Go/NoGo and Alertness from Test of Attentional Performance | Before the 3-week treatment period; 6-month follow up
  Subscales Go/NoGo and Alertness from Test of Attentional Performance; cf. Zimmermann P and Fimm B. Testbatterie zur Aufmerksamkeitsprüfung (TAP). Herzogenrath: PSYTEST Verlag, 2002.
Change in non-verbal episodic memory, as assessed by the Figure Recognition Task from Benton Visual Retention Test | Before the 3-week treatment period; 6-month follow up
  Figure Recognition Task from Benton Visual Retention Test; cf. Benton Sivan A and Spreen O. Benton Test. Bern: Huber, 2009.
Change in mood, as assessed by the German version of the 10-item Stroke Aphasic Depression Questionnaire | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  German version of the 10-item Stroke Aphasic Depression Questionnaire (SADQH-10); cf. Cobley CS, Thomas SA, Lincoln NB, et al. The assessment of low mood in stroke patients with aphasia: reliability and validity of the 10-item Hospital version of the Stroke Aphasic Depression Questionnaire (SADQH-10). Clin Rehabil 2012; 26: 372-381.
Change in health-related quality of life, as assessed by the Stroke and Aphasia Quality of Life Scale | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  Stroke and Aphasia Quality of Life Scale (SAQOL-39g); cf. Hilari K, Lamping DL, Smith SC, et al. Psychometric properties of the Stroke and Aphasia Quality of Life Scale (SAQOL-39) in a generic stroke population. Clin Rehabil 2009; 23: 544-557.
Change in health-related quality of life, as assessed by the EuroQol Health-Related Quality of Life Questionnaire | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  EuroQol Health-Related Quality of Life Questionnaire (EQ-5D-5L); cf. EuroQol G. EuroQol-a new facility for the measurement of health-related quality of life. Health Policy 1990; 16: 199-208.
Change in direct and indirect costs during the 12-month study period, as assessed by the self-developed Patient Resource Consumption Questionnaire | Before the 3-week treatment period; 6- and 12-month follow ups
  Direct and indirect costs during the 12-month study period, as determined by the self-developed Patient Resource Consumption Questionnaire considering common standardized unit cost assumptions.
Change in direct and indirect costs during the 12-month study period, as assessed by the Quality-Adjusted Life Years | Before the 3-week treatment period; 6- and 12-month follow ups
  Quality-Adjusted Life Years; cf. Whitehead SJ and Ali S. Health outcomes in economic evaluation: the QALY and utilities. Br Med Bull 2010; 96: 5-21.
Change in unpaid support provided by family members or friends, as assessed by the Burden of informal caregivers | Before the 3-week treatment period; immediately after the 3-week treatment period; 6- and 12-month follow ups
  Burden of informal caregivers; cf. van Exel NJ, Koopmanschap MA, van den Berg B, et al. Burden of informal caregiving for stroke patients. Identification of caregivers at risk of adverse health effects. Cerebrovasc Dis 2005; 19: 11-17.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof., Principal Investigator — University Medicine Greifswald
Locations (19):
- Germany (19):
  - Aphasiestation RWTH Aachen, Aachen
  - Kliniken Schmieder Allensbach, Allensbach
  - Schön Klinik Bad Aibling Harthausen, Bad Aibling
  - Wicker Klinik Bad Homburg, Bad Homburg
  - Moritz Kliniken Bad Klosterlausnitz, Bad Klosterlausnitz
  - Median Klinik Bad Sülze, Bad Sülze
  - ZAR Berlin, Berlin
  - Kliniken Schmieder Gailingen, Gailingen
  - Klinikum Christophsbad Göppingen, Göppingen
  - University Medicine Greifswald, Department of Neurology, Greifswald
  - BDH-Klinik Greifswald gGmbH, Greifswald
  - Kliniken Schmieder Heidelberg, Heidelberg
  - Hospital zum Heiligen Geist Kempen, Kempen
  - Tagesklinik MPI Leipzig, Leipzig
  - Logo Zentrum Lindlar, Lindlar
  - TheraVent aktiv Marbach, Marbach
  - St. Mauritius Therapieklinik, Meerbusch
  - EUFH Rostock, Rostock
  - Aphasie-Zentrum Vechta gGmbH, Vechta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unger N, Stahl B, Darkow R, Scholz V, Weinmar I, Schmidt J, Breitenstein C, Meinzer M, Grewe T, Floel A. [Transcranial direct current stimulation to enhance training effectiveness in chronic poststroke aphasia-A challenge for recruiting participants]. Nervenarzt. 2024 Apr;95(4):368-375. doi: 10.1007/s00115-023-01572-7. Epub 2024 Jan 4. German. PMID 38175228
- [Derived] Stahl B, Darkow R, von Podewils V, Meinzer M, Grittner U, Reinhold T, Grewe T, Breitenstein C, Floel A. Transcranial Direct Current Stimulation to Enhance Training Effectiveness in Chronic Post-Stroke Aphasia: A Randomized Controlled Trial Protocol. Front Neurol. 2019 Oct 22;10:1089. doi: 10.3389/fneur.2019.01089. eCollection 2019. PMID 31695667